CLINICAL TRIAL: NCT07247110
Title: A Phase 1, Open-Label, Multicenter Study to Assess Safety, Tolerability, Pharmacokinetics, and Efficacy of MK-4716 as Monotherapy and as Part of Combination Therapy in Participants With KRAS-Altered Advanced or Metastatic Solid Tumors
Brief Title: A Clinical Study of MK-4716 in People With Certain Solid Tumors (MK-4716-001)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4716-001; 2025-522495-84 (Registry Identifier: EU CT); U1111-1323-3663 (Registry Identifier: UTN); MK-4701-001 (Other: MSD)
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MK-4716 Dose Escalation (Experimental): Participants receive MK-1084 at varying dose levels and schedules.
  Interventions: Drug: MK-4716
- MK-4716 + Pembrolizumab (Experimental): Participants will receive MK-4716 + Pembrolizumab
  Interventions: Drug: MK-4716; Biological: Pembrolizumab
- MK-4716 + Cetuximab (Experimental): Participants will receive MK-4716 + Cetuximab
  Interventions: Drug: MK-4716; Biological: Cetuximab

INTERVENTIONS:
Drug: MK-4716 — Oral administration
Biological: Pembrolizumab — Intravenous administration
  Other Names: Keytruda
  Arms: MK-4716 + Pembrolizumab
Biological: Cetuximab — Intravenous administration
  Arms: MK-4716 + Cetuximab

SUMMARY:
Researchers are looking for new ways to treat certain advanced or metastatic solid tumors. The goal of this study is to learn about the safety of MK-4716 and if people tolerate it when taken alone or with other treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subset of arm MK-4716 Dose Escalation and subset of arm MK-4716 + Cetuximab: Has a confirmed diagnosis of locally advanced unresectable or metastatic solid tumor
* Subset of arm MK-4716 Dose Escalation and subset of arm MK-4716 + Cetuximab: Must demonstrate presence of Kirsten rat sarcoma viral oncogene homolog (KRAS) alteration
* Subset of arm MK-4716 Dose Escalation and subset of arm MK-4716 + Cetuximab: Has received at least 1 prior line of systemic therapy for locally advanced unresectable or metastatic disease
* Arm MK-4716 + Pembrolizumab: Has a confirmed diagnosis of metastatic non-small cell lung cancer
* Arm MK-4716 + Pembrolizumab: Must demonstrate presence of KRAS alteration
* Arm MK-4716 + Pembrolizumab: Must be untreated
* Arm MK-4716 + Cetuximab: Must be eligible for cetuximab
* Has measurable disease
* Has the ability to swallow and retain oral medication

Exclusion Criteria:

* Arm MK-4716 + Pembrolizumab: Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Arm MK-4716 + Pembrolizumab: Has received any prior immunotherapy and was discontinued from that treatment
* Arm MK-4716 + Pembrolizumab: Has active autoimmune disease that has required systemic treatment in the past 2 years. Hormonal supplementation (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed
* History of human immunodeficiency virus infection
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has a known active central nervous system metastases and/or carcinomatous meningitis
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has Hepatitis B or Hepatitis C virus infection
* History of stem cell/solid organ transplant
* Has not adequately recovered from major surgery or has ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience One or More Dose-Limiting Toxicities (DLT) | Up to approximately 28 days
  A DLT is defined as the occurrence of protocol-specified toxicities, unless clearly related to disease progression or intercurrent illness.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of MK-4716 | At designated timepoints (up to approximately 58 days)
  Blood samples will be collected to determine the AUC of MK-4716.
Maximum Plasma Concentration (Cmax) of MK-4716 | At designated timepoints (up to approximately 58 days)
  Blood samples will be collected to estimate Cmax of MK-4716.
Trough Plasma Concentration (Ctrough) of MK-4716 | At designated timepoints (up to approximately 19 months)
  Blood samples will be collected to determine the Ctrough of MK-4716.
Half-Life (t1/2) of MK-4716 | At designated timepoints (up to approximately 58 days)
  Blood samples will be collected to determine the t1/2 of MK-4716.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- United States (2):
  - NEXT Oncology ( Site 0051), Irving, Texas
  - NEXT Virginia ( Site 0054), Fairfax, Virginia
- Israel (3):
  - Rambam Health Care Campus ( Site 0252), Haifa
  - Rabin Medical Center ( Site 0253), Petah Tikva
  - Sheba Medical Center ( Site 0251), Ramat Gan
- Spain (2):
  - Hospital Clinic de Barcelona ( Site 0362), Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 0361), Madrid

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/